CLINICAL TRIAL: NCT02940639
Title: A National, Prospective, Non-Interventional Study (NIS) in Patients With Advanced/Metastatic Renal Cell Carcinoma Starting 1st Line Nivolumab and Ipilimumab Combination Therapy or Nivolumab Monotherapy After Prior Therapy
Brief Title: Real-Life Effectiveness and Safety in Participants With Advanced/Metastatic Renal Cell Carcinoma Starting 1st Line Nivolumab and Ipilimumab Combination Therapy or Nivolumab Monotherapy After Prior Therapy
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA209-653
Record Dates: First submitted 2016-10-12; First posted 2016-10-21 (Estimated); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cohort 1: Participants with advanced/metastatic renal cell cancer (RCC) starting nivolumab monotherapy after prior therapy
- Cohort 2: Participants with advanced/metastatic RCC starting 1st line therapy with nivolumab and ipilimumab combination therapy, in intermediate/poor risk participants

SUMMARY:
The purpose of this study is to estimate overall survival over a 5-year follow-up period among adult participants with advanced/metastatic kidney cancer, starting 1st line nivolumab and ipilimumab combination therapy or nivolumab monotherapy after prior therapy, in real-life conditions in Germany

ELIGIBILITY:
Inclusion Criteria:

Adult participants, at least 18 years of age at time of treatment decision

* Diagnosis of advanced/metastatic renal cell carcinoma (RCC) (confirmed by histology or cytology)
* Treatment decision to initiate a treatment with nivolumab and ipilimumab or nivolumab for the first time for the treatment of advanced/metastatic RCC (according to the label approved in Germany) has already been taken
* Signed informed consent

Exclusion Criteria:

* Participants with a diagnosis of a cancer other than advanced/metastatic advanced RCC within the past five years, ie, a cancer other than advanced/metastatic RCC that requires systemic or other treatment. Participants that have been treated curatively more than five years ago with no evidence of recurrence and prostate cancer patients in active surveillance can be included.
* Participants previously treated with nivolumab and/or ipilimumab
* Participants currently included in an interventional clinical trial for their locally advanced or metastatic RCC. Participants who have completed their participation in an interventional trial; or who are not receiving study drug anymore and who are only followed-up for OS can be enrolled.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants who are at least 18 years of age at the time of the treatment decision with the diagnosis of advanced/metastatic RCC (histologically or cytologically confirmed) and whose physician has already decided to initiate a treatment with 1st line nivolumab and ipilimumab nivolumab combination therapy in intermediate/poor risk participants according to International Metastatic RCC Database Consortium (IMDC) score or with nivolumab monotherapy after prior therapy for the first time for the treatment of advanced/metastatic RCC, according to the label approved in Germany.
Sampling Method: Probability Sample
Enrollment: 499 (Actual)
Dates: Start 2016-10-27 (Actual); Primary Completion 2025-06-03 (Actual); Study Completion 2025-06-03 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) | Approximately 5 years
  In participants with nivolumab and ipilimumab or nivolumab therapy

SECONDARY OUTCOMES:
Overall Survival (OS) | Approximately 5 years
  Separate by nivolumab and ipilimumab or nivolumab therapy, estimated overall lines of therapy, per line of therapy, per cohort, per index date (initial diagnosis vs start of therapy in the trial) and per subgroups of interest.
Progression-Free Survival (PFS) | Approximately 5 years
Overall response rate (ORR) | Approximately 5 years
Best Overall Response (BOR) | Approximately 5 years
Best Overall Response Rate (BORR) | Approximately 5 years
Duration of Response | Approximately 5 years
Distribution of socio-demographic characteristics | Approximately 5 years
  Socio-demographic characteristics (Gender, Height, Weight, Age) will be summarized using descriptive statistics.
Distribution of clinical characteristics | Approximately 5 years
  Clinical characteristics (Initial Diagnosis of RCC, Histological subtypes, Performance status, Comorbidities, history of cancer) will be summarized using descriptive statistics
Distribution of Renal Cell Carcinoma (RCC) Treatment History | At Baseline
Distribution of Nivolumab Treatment Characteristics | At initiation - index date, baseline
  Nivolumab monotherapy (cohort 1) or nivolumab and ipilimumab combination therapy (cohort 2)
Distribution of Treatment Patterns | Approximately 5 years
  Details on prior and evolution of current treatment patterns
Incidence rate of Adverse Events (AEs), treatment-related AEs, select AEs and other immune-related AEs | Approximately 5 years
Distribution of Adverse Events (AE) characteristics | Approximately 5 years
Distribution of severity of Adverse Events (AEs) | Approximately 5 years
Distribution of management of Adverse Events (AEs) | Approximately 5 years
Quality of Life as assessed by Functional Assessment of Cancer Therapy - Kidney Symptom Index (FKSI-19) Questionnaire | Approximately 5 years
Utility as assessed by European Quality of Life-5 Dimensions (EQ-5D) Questionnaire | Approximately 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution - 0001, Jena, Germany

REFERENCES:
- [Derived] Bedke J, Grimm MO, Grunwald V. Collection of real-world data on nivolumab's effectiveness in renal cell carcinoma: rationale for an observational study. Future Oncol. 2018 May;14(11):1023-1034. doi: 10.2217/fon-2017-0637. Epub 2018 Jan 12. PMID 29325434
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html